CLINICAL TRIAL: NCT02443792
Title: Adult Male Circumcision With Unicirc Under Topical Anesthetic vs Open Surgical Circumcision: a Randomized Controlled Trial
Brief Title: Unicirc vs Open Surgical Circumcision
Acronym: Unicirc004
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Simunye Primary Health Care (Other)
Responsible Party: Principal Investigator, Justin Shenje, MB ChB, PI, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Unicirc004
Record Dates: First submitted 2015-04-10; First posted 2015-05-14 (Estimated); Results first posted 2016-01-20 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2018-09

CONDITIONS: Circumcision, Male
MeSH Terms: interventions — Tissue Adhesives; Conversion to Open Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Unicirc with tissue adhesive (Experimental): Unicirc under topical anesthetic w/ cyanoacrylate wound sealing
  Interventions: Procedure: Unicirc with tissue adhesive
- Open Surgical (Active Comparator): Open surgical circumcision under local anesthetic with suturing
  Interventions: Procedure: Open Surgical

INTERVENTIONS:
Procedure: Unicirc with tissue adhesive — As above
  Arms: Unicirc with tissue adhesive
Procedure: Open Surgical — As above
  Arms: Open Surgical

SUMMARY:
RCT of Unicirc under topical anesthetic w/ cyanoacrylate wound sealing vs. open surgical circumcision under local anesthetic with suturing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male
* Uncircumcised
* With normal penile anatomy

Exclusion Criteria:

* Concurrent illness
* History of bleeding disorder
* Past reaction to local anesthetic
* Infection
* Penile abnormality which could complicate circumcision

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2015-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Lonmin Hospital, Marikana, Northwest, South Africa

REFERENCES:
- [Background] Millard PS, Goldstuck ND. No-needle, single-visit adult male circumcision with Unicirc: a multi-centre field trial. PLoS One. 2015 Mar 30;10(3):e0121686. doi: 10.1371/journal.pone.0121686. eCollection 2015. PMID 25822727
- [Derived] Shenje J, Millard PS. Sutureless Adult Voluntary Male Circumcision with Topical Anesthetic: A Randomized Field Trial of Unicirc, a Single-Use Surgical Instrument. PLoS One. 2016 Jun 14;11(6):e0157065. doi: 10.1371/journal.pone.0157065. eCollection 2016. PMID 27299735

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Unicirc With Tissue Adhesive | Open Surgical
Started | 50 | 25
Completed | 43 | 23
Not Completed | 7 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Unicirc With Tissue Adhesive | Open Surgical | Total
Number analyzed (Participants) | 50 | 25 | 75
Age, Customized [Number; unit: participants]
  Age 18-25 | 3 | 2 | 5
  Age 26-35 | 19 | 12 | 31
  Age 36+ | 28 | 11 | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 50 | 25 | 75
Region of Enrollment [Number; unit: participants]
  South Africa | 50 | 25 | 75

OUTCOME MEASURES:

1. Primary Outcome: Time Elapsed From First Clamp (Surgical) or Start of Insertion of Bell (Unicirc) to Beginning of Wound Dressing
Description: Time elapsed from first clamp (surgical) or start of insertion of bell (Unicirc) to beginning of wound dressing
Time Frame: Up to 30 minutes
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Unicirc With Tissue Adhesive | Open Surgical
Number analyzed (Participants) | 50 | 25
Minutes | 12 [11 to 17] | 25 [21 to 35]

2. Secondary Outcome: Surgical Pain 0=no Pain; 10=Worst Pain Ever
Description: Self-described pain severity during procedure (scale 1 to 10). 0=no pain, 5=moderate pain, 10=worst pain ever
Time Frame: Up to 30 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Unicirc With Tissue Adhesive | Open Surgical
Number analyzed (Participants) | 50 | 25
units on a scale | 1.7 (1.3) | 1.9 (2.4)

3. Secondary Outcome: Completely Healed at 4 Weeks
Description: Number of participants who were completely healed at 4 weeks
Time Frame: At the 4-week followup visit
Measure: Number; unit: participants
Arm/Group | Unicirc With Tissue Adhesive | Open Surgical
Number analyzed (Participants) | 50 | 25
participants | 39 | 16

4. Secondary Outcome: Wound Dehiscence
Description: Proportion experiencing wound dehiscence (< 2 cm vs > 2 cm)
Time Frame: Up to 4 weeks
Measure: Number; unit: participants
Arm/Group | Unicirc With Tissue Adhesive | Open Surgical
Number analyzed (Participants) | 50 | 25
participants
  Dehiscence > 2 cm longitudinally | 0 | 0
  Dehiscence < 2 cm longitudinally | 14 | 4

5. Secondary Outcome: Infection
Description: Proportion experiencing post-op infection, determined clinically (treated with antibiotics)
Time Frame: Up to 4 weeks
Measure: Number; unit: participants
Arm/Group | Unicirc With Tissue Adhesive | Open Surgical
Number analyzed (Participants) | 50 | 25
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Any any time during study (4-6 weeks)
Arm/Group | Unicirc With Tissue Adhesive | Open Surgical
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/25
Other Adverse Events (participants affected / at risk) | 3/50 | 0/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Unicirc With Tissue Adhesive (N=50) | Open Surgical (N=25)
Post-op bleeding (Surgical and medical procedures) | 1 (1) | 0 (0) — Bleeding requiring sutures
Intraoperative bleeding requiring sutures (Surgical and medical procedures) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No